CLINICAL TRIAL: NCT04007471
Title: Adolescent Dysmenorrhea : Prevalence, Severity, Experience and Management in the Use of Medication in High School Girls in Ille-et-Vilaine
Acronym: DAPsvs
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC19_30017_DAPsvs
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2019-07

CONDITIONS: Adolescent Dysmenorrhea
Keywords: Dysmenorrhea; Primary dysmenorrhea; Secondary dysmenorrhea; Pelvic pain; Menstrual pain; Adolescent; Endometriosis
MeSH Terms: conditions — Dysmenorrhea; Pelvic Pain; Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Anonymous survey — Anonymous questionnaire to determine the prevalence of dysmenorrhea of adolescent girls, to assess the severity of dysmenorrhea, how girls experience their menses, the consequences on daily living activities or at school, and how they manage their pain.

SUMMARY:
Dysmenorrhea or painful menstruation is a common symptom of menses. Dysmenorrhea is defined as a painful, cramping sensation in the lower abdomen or back associated with menstrual periods and is classified into primary and secondary types. Primary dysmenorrhea is painful menstrual periods not due to other diseases, and often occurs soon after menarche. Secondary dysmenorrhea is due to an underlying pelvic abnormality, such as endometriosis.

Dysmenorrhea is the most common gynecological complaint. In many studies, the prevalence of primary dysmenorrhea varies between 34 % in 2010 in Egypt, 86.6% in 2002 in Switzerland, and 21% in 1999 in France.

Nowadays, physiopathology is better understood, which suggests that the investigators have treatments Although dysmenorrhea is a common concern, many women never seek medical advice, even though treatments are easily available and simple.

In fact, despite the high prevalence, dysmenorrhea is undertreated and even disregarded by health professionals, and the girls themselves, who may accept it as a normal part of the menstrual cycle.

The pain occurs just before and/or during menstruation ; it can be mild to severe and is frequently associated with many other symptoms, like nausea, vomiting, headache, diarrhea, tiredness and has many consequences in wellbeing and school. Dysmenorrhea is known to be the first cause of absenteism from school, and appears to have many consequences and a real impact on women's daily activities, which is why it's a public health problem.

Because of the lack of recent studies in France, the aim of this study is to evaluate the prevalence of adolescent dysmenorrhea. The investigators also assessed its severity, how adolescent girls experienced their menses, and how they manage their pain (seeking medical consultation, use of medication).

The investigators used a self-assessment questionnaire in a cohort of high school girls, aged 15 to 19 years old, during April and May of 2019, in 8 private and public high schools in Ille-et-Vilaine.

DETAILED DESCRIPTION:
It was an observational, quantitative and prospective study, in a cohort of adolescent girls, to assess the prevalence of adolescent dysmenorrhea through an anonymous self-assessment questionnaire, which took place in 8 randomised public and private high schools in Ille-et-Vilaine, Brittany, France.

Only adolescents aged between 15 and 19 years old who agreed to participate were included. Girls who had experienced primary or secondary amenorrhea for more than 6 months in the past year were excluded.

The target number of participants was 770 adolescents girls aged between 15 and 19 years old.

The main objective was to determine the prevalence of dysmenorrhea within adolescent girls in a sample in France.

The other objectives were to assess the severity, how girls experienced their menses, the consequences on daily living activities or at school, and how they manage their pain.

The severity of dysmenorrhea were assessed with Andersch and Milsom's scale and Numerical Rating Scale (NRS).

First of all, the investigators also obtained the authorization of the Committee of Protection of People of Montpellier University Hospital.

After that, the investigators contacted the high school principals of the 8 high schools which were randomized, and obtained their authorization to organise this study in their schools.

The investigators gave an information to the parents and adolescent girls about ten days before the study. If a girl or their parents didn't want their daughter to participate, they could inform the high school principal or the school nurse. The investigators asked the nurse or the directos of high schools to make a randomisation of the girls.

Then, the investigators gathered them in a classroom, with no boys, to make sure that the girls felt free and confident enough to complete the questionnaire in the most honest way. The investigators gave them the questionnaires, and let them complete it, which took about 15-20 minutes.

The main investigator was present to answer the girls if any questions were not understood.

After completion, the questionnaires were immediately retrieved by the main investigator.

Finally, the investigators briefly communicated what menses are and other symptoms, how to relieve the pain, with or without medication, and in what case the girls must see a doctor. The investigators gave them an advice sheet. The aim was to improve the management of dysmenorrhea and their quality of life by informing adolescent girls of the availability of effective therapy and the need to consult a doctor in some situations.

A sample of 960 adolescents completed the questionnaire, and 19 were excluded. The prevalence of dysmenorrhea will be calculated. Then, the investigators will analyze the sample.

These results will provide a better understanding of dysmenorrhea, its recent prevalence, its severity, its influencing factors and its consequences on daily activities. This study will help to better know the impact of dysmenorrhea, which is frequently underestimated and misunderstood by girls themselves, their parents, their families and their teachers.

In addition, throughout this study, the reasons why adolescent girls may not want to seek medical consultation might be known. The investigators could as general practitionner or gynecologist better explain and advise adolescent girls, offer them relief and better conditions of life, while staying aware of the possibility of secondary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent girls aged between 15 and 19 years old
* Menstruating adolescent girls
* Accept participation
* Schooled in one of the 8 randomised public and private high schools in Ille-et-Vilaine

Exclusion Criteria:

* Girls under 15 or over 19 years old
* If a girl or their parents didn't want their daughter to participate
* Primary or secondary amenorrhea during more than 6 months in the past year

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Cohort of adolescent girls aged between 15 and 19 years old who go to a private or public highschool in Ille-et-Vilaine A sample of 960 girls were obtained
Sampling Method: Probability Sample
Enrollment: 979 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
Prevalence of dysmenorrhea | Inclusion day
  " During last past year, have you ever experienced pain in your lower abdomen or back associated with menstrual periods ? " " Never " - " Sometimes " - " Always "

CONTACTS AND LOCATIONS:
Overall Officials: Maud BIDET, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France